CLINICAL TRIAL: NCT06894563
Title: On the Move: Center and Home-Based Exercise to Enhance Mobility in Diabetic Foot Ulcer Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HP-00113990
Record Dates: First submitted 2025-03-07; First posted 2025-03-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: Clinical trial; Mobility; Diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, outcome assessor blinded, parallel group clinical trial comparing a 12-week exercise regimen to standard of care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12-week exercise regimen (Experimental): Consistent with current physical activity recommendations for older adults, participants randomized in this arm will be prescribed 5 days/week of exercise, with seated cycling exercise performed on 3 days a week and strength/balance exercise performed 2 days a week.
  Interventions: Behavioral: 12-week exercise regimen
- 12-week standard of care (Placebo Comparator): Participants in this group will be provided with guidance on the current standard of care. This includes guidance that these patients should slowly increase ambulation with appropriately fitted footwear.
  Interventions: Behavioral: 12-week standard of care

INTERVENTIONS:
Behavioral: 12-week exercise regimen — Consistent with current physical activity recommendations for older adults, participants randomized in this arm will be prescribed 5 days/week of exercise, with seated cycling exercise performed on 3 days a week, and strength/balance exercise performed 2 days a week.
  Arms: 12-week exercise regimen
Behavioral: 12-week standard of care — Participants in this group will be provided with guidance on the current standard of care. This includes guidance that these patients should slowly increase ambulation with appropriately fitted footwear.
  Arms: 12-week standard of care

SUMMARY:
Foot ulcers and amputations are a common and feared complication for people with diabetes. People with a diabetic foot ulcer have a higher risk of dying within five years than people with diabetes without an ulcer. At least one in four people with a new diabetic foot ulcer will die within five years, largely due to cardiovascular causes. The reasons for this increased mortality involve decreased mobility.

People with a recently healed diabetic foot ulcer are considered "in remission" as opposed to "cured" because the underlying medical problems (e.g., peripheral neuropathy, peripheral arterial disease) which led to their ulcer are still present. Once in remission, the current standard of care is to slowly increase ambulation with appropriate footwear so as not to promote ulcer recurrence. The problem is that people rarely return to the recommended level of mobility. The ability to safely maintain mobility with aging is critical, as immobility is the leading cause of nursing home admissions.

This is a clinical trial to test the feasibility and acceptability of an exercise regimen that transitions from in-person to home-based. The investigators will also assess if this exercise regimen can increase mobility and function without increasing diabetic foot ulcer recurrence by improving mobility, lower extremity strength, lower extremity tissue perfusion and glycemic control.

DETAILED DESCRIPTION:
Population: 60 Veterans with a healed foot ulcer in the last 3-15 months

Site: VA Maryland Health Care System (VAMHCS)

Study Duration: Approximately 3 years

Study Design: Randomized, outcome assessor blinded, clinical trial comparing a) a 12-week exercise regimen to b) standard of care

Objectives:

Primary: To assess the feasibility and acceptability of the intervention and estimate the effect of the intervention on 6-minute walk distance.

Secondary:

The effect of the intervention on other measures of mobility and function including gait speed, the Modified Physical Performance Test, steps per day and community mobility following the 12-week intervention and 6-months after to assess retention of the intervention.

The effect of the intervention on lower extremity strength, perfusion of the foot and glycemic control.

Treatment Regimens: 12-week exercise regimen to standard of care

Duration of Participant's Participation: Up to 10 months

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 50 years
* Diagnosis of diabetes
* Plantar foot ulcer which healed within the last 3-15 months
* Two feet (can have healed minor amputations of fore and midfoot)
* Willing to wear appropriately fitted footwear for exercise regimen
* Ambulatory without walker
* Willing to enroll in the PODIMETRICS SmartMat program
* Able to give written informed consent

Exclusion Criteria:

* Unable to perform the exercise interventions (e.g. due to hearing or visual impairment)
* Anticipated foot surgery in the next 4 months
* Participating in another exercise program
* Severe peripheral arterial disease (Fontaine stage 3 rest pain or 4 ischemic ulcers/gangrene)
* Current plantar foot ulcer
* Any other criteria which, in the investigator's opinion, would compromise the ability of a subject to participate safely

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walk distance | 12 weeks
  Using standard procedures participants will be asked to walk as far as possible in 6 minutes along a 100-foot course. Primary clinical outcome is total distance covered.

SECONDARY OUTCOMES:
Acceptability and Feasibility | 12 weeks
  Acceptability and feasibility of the intervention by the participant will be measured using the Usage Rating Profile-Intervention (URPI) at each phase or transition of the intervention and through a semi-structured interview.
Adherence to the exercise regimen | 12 weeks
  Adherence to the exercise regimen will be assessed using written logs of attendance to group exercise.
SmartMat metrics | 12 weeks
  Use of SmartMat to measure the temperature of the plantar aspect of the foot and triggers (sustained asymmetric increase in temperature) for a potential foot complication.
Community Mobility | 12 weeks
  Community mobility will be assessed using the Life-Space Assessment (LSA).
Mobility Function | 12 weeks
  Mobility function will be assessed using the Modified Physical Performance Test (MPPT)
Physical Activity | 12 weeks
  Physical activity will be assessed as average steps per day, measured with a FitBit.
Muscular strength | 12 weeks
  Knee extension and plantar flexion strength will be assessed using a MicroFET 2 Handheld Dynamometer.
Perfusion | 12 weeks
  Cutaneous perfusion will be assessed on the dorsal and plantar surfaces of the foot using laser Doppler flowmetry using the PeriFlux System 5000.
Glycemic Control | 12 weeks
  Blood samples will be obtained by venipuncture for HbA1c measurement.

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA. A limited dataset will be created and shared pursuant to a Data Use Agreement. Final data sets will be maintained locally until enterprise-level resources become available. Upon request, we will provide an electronic limited dataset to others in the scientific community with the implementation of appropriate data use agreements.
Supporting Information: Study Protocol, SAP
Access Criteria: Implementation of appropriate data use agreements. Email the study PI, Dr. Mary-Claire Roghmann (mroghmann@som.umaryland.edu), to start the process.